CLINICAL TRIAL: NCT05672511
Title: The Effect of Simulation Teaching Method on Midwifery Students' Knowledge and Skills of Vaginal Examination in Labor: A Randomized Controlled Study
Brief Title: The Effect of Simulation Teaching Method on Midwifery Students'
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Döndü BATKIN ERTÜRK, Assistant Proffesor Dr, Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: TOKAT01
Record Dates: First submitted 2023-01-03; First posted 2023-01-05 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Educational Problems
Keywords: Vaginal Examination; Knowledge; Skill; Simulation; Teaching

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervention group (Experimental): Randomly determined experimental group students will perform eight vaginal examination scenarios different in terms of cervical effacement, cervical dilatation, presence of amniotic membrane, presenting fetus part, position of the fetus and fetal descent on the fetal monitoring and labor progress model set in the laboratory.
  Interventions: Behavioral: Simulation Teaching Method
- Control group (No Intervention): . The control group will not receive any simulation training

INTERVENTIONS:
Behavioral: Simulation Teaching Method — Randomly determined experimental group students will perform eight vaginal examination scenarios different in terms of cervical effacement, cervical dilatation, presence of amniotic membrane, presenting fetus part, position of the fetus and fetal descent on the fetal monitoring and labor progress model set in the laboratory. The control group will not receive any simulation training. Both groups will be given a knowledge test after teaching with simulation. Students in both groups will fill out a form evaluating their skills in performing the steps of vaginal examination before each vaginal examination is performed on women in the clinic.
  Arms: İntervention group

SUMMARY:
This study was planned to evaluate the effect of simulation teaching method on the knowledge and skills of midwifery students in applying vaginal examination in labor.The study was planned as a randomized controlled trial.Research Tokat It will be held between 10.10.2022 and 10.06.2023 at Gaziosmanpaşa University Faculty of Health Sciences, Tokat Gaziosmanpaşa University Health Research and Application Hospital and Tokat Provincial Health Directorate Tokat State Hospital.The population of the research will consist of students (N=102) who are students of Tokat Gaziosmanpaşa University Health Sciences Faculty Midwifery Department, who took the Normal Birth and Postpartum Period course for the first time in the 2022-2023 academic year, and who have not had a vaginal examination before. The sample of the randomized controlled study was calculated in the G*Power 3.1 program . Accordingly, the number of samples to be included in the study for an error margin of 0.05 with a statistical power of 80% was calculated as n= 51 for the experimental group and n= 51 for the control group for each group.The Effect of Simulation Teaching Method on Midwifery Students' Knowledge and Skills of Applying Vaginal Examination in Labor: The Randomized Controlled Study Questionnaire consists of four parts.Randomly determined experimental group students will perform eight vaginal examination scenarios different in terms of cervical effacement, cervical dilatation, presence of amniotic membrane, presenting fetus part, position of the fetus and fetal descent on the fetal monitoring and labor progress model set in the laboratory. The control group will not receive any simulation training.

DETAILED DESCRIPTION:
Two skills, abdominal palpation and vaginal examination, are used to clinically monitor the progress of labor. Vaginal examination is the most accepted method of measuring the progress of labor. Vaginal examination, which is routinely applied in the evaluation of the progress of labor, is an important part of midwifery care. However, the accuracy level of vaginal examination for new students is reported to be low. This basic skill is appropriate for women in labor a learned tactile/tactile one that requires consistency to manage is skill. Therefore, it cannot be learned through observation alone; In order to acquire this skill, students must perform a large number of vaginal examinations in women who have given birth. The usual/classic training technique for teaching vaginal examination is that the midwifery student performs the vaginal examination on the woman in labor under the supervision of an experienced obstetrician, then the experienced obstetrician repeats this examination to determine the accuracy of the trainee student's assessment.

Teaching method with simulation models is very important in learning this basic midwifery skill. Simulation is a teaching and learning method that creates an artificial or theoretical experience, engaging the student in an activity that reflects real-life conditions without the risk-taking consequences of real conditions. In other words, it is a teaching approach based on a model developed in accordance with reality to support learning. Simulation is actually ethical in order not to harm the patient in practice is a must. Simulation-based learning improves the understanding, retention and active use of knowledge and skills, reduces the student's pre-application anxiety, and increases self-confidence. It is seen that simulation, which has been widely used in medical education in recent years, is also used as a teaching method in the development of practice skills of midwifery students. There are several studies in the literature evaluating the effect of simulation training on students' vaginal examination skills. Teaching obstetric vaginal examination techniques to medical students conducted to evaluate the benefits of simulation training vaginal examination of students receiving simulation training in a study accuracy is important according to students who did not receive simulation training was found to be high. In this study, it was concluded that simulation training helped inexperienced students improve their vaginal examination skills before performing such procedures on real patients. In the study of Abbas et al. (2019), interns who performed simulated examination showed significantly higher accuracy in vaginal examination evaluations than the control group. This study was planned to evaluate the effect of simulation teaching method on the knowledge and skills of vaginal examination in labor in midwifery students.

Type of Study: The study was planned as a randomized controlled trial.

Place and Time of the Research: The research will be carried out at Tokat Gaziosmanpaşa University Faculty of Health Sciences, Tokat Gaziosmanpaşa University Health Research and Application Hospital and Tokat Provincial Health Directorate Tokat State Hospital between 10.10.2022-10.06.2023.

Research Tokat It will be held between 10.10.2022 and 10.06.2023 at Gaziosmanpaşa University Faculty of Health Sciences, Tokat Gaziosmanpaşa University Health Research and Application Hospital and Tokat Provincial Health Directorate Tokat State Hospital.

Population and Sample of the Research:

The population of the research will consist of students (N=102) who are students of Tokat Gaziosmanpaşa University Health Sciences Faculty Midwifery Department, who took the Normal Birth and Postpartum Period course for the first time in the 2022-2023 academic year, and who have not had a vaginal examination before. The sample of the randomized controlled study was calculated in the G*Power 3.1 program . Accordingly, the number of samples to be included in the study for an error margin of 0.05 with a statistical power of 80% was calculated as n= 51 for the experimental group and n= 51 for the control group for each group. Students will be assigned to the groups by adding them to the first column of the Microsoft Excel program according to the sequence number in the list and deriving the number in the second column.

Data Collection Tools The Effect of Simulation Teaching Method on Midwifery Students' Knowledge and Skills of Applying Vaginal Examination in Labor: The Randomized Controlled Study Questionnaire consists of four parts.

A. Socio-demographic characteristics of students There are 16 questions in total in this section. Midwifery students' age, marital status, graduated school, family structure, place of residence, education level of mother and father, perception of income status, place of residence of the family, the presence of health personnel in the family members, their duties, if any, satisfaction with the midwifery department, order of preference for the midwifery profession, overall academic grade point average, the relationship between finding the theoretical knowledge and skills sufficient in applying vaginal examination B. List of skills for students to perform vaginal examination practice steps This is the section where the skills of the students in performing the vaginal examination application steps (22 items) prepared by the researchers by examining the literature are evaluated. The items will be evaluated by the researchers as they did or did not. The first vaginal examination on the woman in the clinic will be filled in both groups before the application.

C. Vaginal examination evaluation results of the students in the clinic This is the section where the evaluation results of the midwifery student and experienced health professional (cervical effacement, cervical dilatation, presence of amniotic membrane, presenting fetus part, position of the fetus and fetal descent) will be recorded in the vaginal examinations performed on women in the clinic for both groups.

D. Vaginal Examination Knowledge Test It is a knowledge test for the vaginal examination application prepared by the researchers by examining the literature. It consists of 12 questions. A total knowledge score will be obtained by calculating the points given as 1 point for the correct answer and 0 for the wrong answer for each multiple-choice question. It will be done to both groups after teaching with simulation and after the completion of the vaginal examinations on the woman in the clinic.

Application of the Research:

All students who take the Normal Birth and Postpartum Term course will be given a theoretical course on the steps of vaginal examination in labor and the criteria to be evaluated in vaginal examination. Informed consent will be obtained from all students who voluntarily agree to participate in the study after being informed about the study. Students will be asked to fill in a questionnaire prepared by the researchers examining the socio-demographic characteristics of the students. Randomly determined experimental group students will perform eight vaginal examination scenarios different in terms of cervical effacement, cervical dilatation, presence of amniotic membrane, presenting fetus part, position of the fetus and fetal descent on the fetal monitoring and labor progress model set in the laboratory. The control group will not receive any simulation training. Both groups will be given a knowledge test after teaching with simulation. Students in both groups will fill out a form evaluating their skills in performing the steps of vaginal examination before each vaginal examination is performed on women in the clinic. For both groups, vaginal examination evaluation results (cervical effacement, cervical dilatation, presence of amniotic membrane, presenting fetus part and fetal descent) of midwifery student and experienced health professional (midwife, nurse and doctor) will be recorded in four vaginal examinations performed on women in the clinic. In this study, the vaginal examination procedure normally used by midwifery students during their professional practice in health institutions will be used. An experienced health professional will perform the vaginal examination in the woman in labor, and then the midwifery student will repeat the vaginal examination on the same woman under the supervision of an experienced health professional and the evaluation findings will be compared. Informed consent will be obtained from women prior to the vaginal examination, infection control measures will be taken during the examinations (hand washing, wearing sterile gloves and avoiding frequent vaginal examinations), and women's privacy will be respected as much as possible. The findings of experienced health professionals will be accepted as the gold standard in the study. Student findings compatible with the findings of the experienced healthcare professional will be evaluated as correct, and student findings that are not compatible with or could not be evaluated with the findings of the experienced healthcare professional will be evaluated as incorrect. After the completion of the vaginal examinations on the woman in the clinic, the knowledge test will be performed for the second time in both groups. When the research data is completed, all students in the control group will have applications on the fetal monitoring and labor progress model set by the simulation teaching method, in order to ensure equality of opportunity in education, by the researchers.

LIST OF PARAMETERS TO BE USED IN THE RESEARCH

* Assessment of students' ability to perform vaginal examination application steps
* Vaginal examination evaluation parameters (cervical effacement, cervical dilatation, presence of amniotic membrane, presenting fetus part and fetal descent)
* Knowledge test for vaginal examination

ELIGIBILITY:
Inclusion Criteria:

* who took the Normal Birth and Postpartum Period course for the first time in the 2022-2023 academic year, and who have not had a vaginal examination before.

Exclusion Criteria:

* Those who have done 5 or more vaginal examinations on real pregnant women before.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
List of skills for students to perform vaginal examination practice steps | baseline
  This is the section where the skills of the students in performing the vaginal examination application steps (22 items) prepared by the researchers by examining the literature are evaluated. The items will be evaluated by the researchers as they did or did not. The first vaginal examination on the woman in the clinic will be filled in both groups before the application.

CONTACTS AND LOCATIONS:
Overall Officials: Döndü BATKIN ERTÜRK, Study Director — Midwifery
Locations (1):
- Tokat Gaziosmanpasa University, Faculty of Health Sciences, Midwifery Department, Tokat Province, Turkey/Tokat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pratinidhi, A., Patange, R., Patil, S., Salunkhe, J., & Samson, S. (2014). Testing of simulation training device for assessment of cervical dilatation among nursing student of Karad, India
- [Background] Muliira RS, Seshan V, Ramasubramaniam S. Improving vaginal examinations performed by midwives. Sultan Qaboos Univ Med J. 2013 Aug;13(3):442-9. Epub 2013 Jun 25. PMID 23984031
- [Background] Huhn KA, Brost BC. Accuracy of simulated cervical dilation and effacement measurements among practitioners. Am J Obstet Gynecol. 2004 Nov;191(5):1797-9. doi: 10.1016/j.ajog.2004.07.062. PMID 15547567
- [Background] Arias T, Tran A, Breaud J, Fournier JP, Bongain A, Delotte J. A prospective study into the benefits of simulation training in teaching obstetric vaginal examination. Int J Gynaecol Obstet. 2016 Jun;133(3):380-4. doi: 10.1016/j.ijgo.2015.08.028. Epub 2016 Feb 23. PMID 26971257
- [Background] Chahine, E. B., Rizk, S., Young, M., Moynihan, A., Arluck, J., & Walker, P. (2018). Intern Bootcamp Cervical Dilation Simulation: Findings and Assessment [34M]. Obstetrics & Gynecology, 131, 150S.
- [Background] Roosevelt L, Diebel M, Zielinski RE. Achieving competency in vaginal examinations: The challenge of balancing student learning needs with best practice in maternity care. Midwifery. 2018 Jun;61:39-41. doi: 10.1016/j.midw.2018.02.016. Epub 2018 Feb 23. PMID 29524775
- [Background] Cass GK, Crofts JF, Draycott TJ. The use of simulation to teach clinical skills in obstetrics. Semin Perinatol. 2011 Apr;35(2):68-73. doi: 10.1053/j.semperi.2011.01.005. PMID 21440813
- [Background] Bastable, S. B. (2017). Nurse as educator: Principles of teaching and learning for nursing practice. jones & bartlett learning.
- [Background] Aslan, M. Günay, O. Çetinkaya, F. Mazıcıoğlu, M., (2002). Tıp Eğiticileri İçin Eğitim Becerileri Rehberi. Erciyes Üniversitesi Tıp Fakültesi, Yayın No:70, 80-88, Kayseri.
- [Background] McEwen BS, Sapolsky RM. Stress and cognitive function. Curr Opin Neurobiol. 1995 Apr;5(2):205-16. doi: 10.1016/0959-4388(95)80028-x. PMID 7620309
- [Background] Nitsche JF, Shumard KM, Fino NF, Denney JM, Quinn KH, Bailey JC, Jijon R, Huang C, Kesty K, Whitecar PW, Grandis AS, Brost BC. Effectiveness of Labor Cervical Examination Simulation in Medical Student Education. Obstet Gynecol. 2015 Oct;126 Suppl 4:13S-20S. doi: 10.1097/AOG.0000000000001027. PMID 26375554
- [Background] Driscoll, Mp., (2005). Pyschology of Learning for İnstruction, 3rd Ed. New York: Pearson.
- [Background] Tiffen, J. Graf, N. Corbridge, S., (2009). Effectiveness of a Low-Fidelity Simulation Experience in Building Confidence Among Advanced Practice Nursing Graduate Students. Clinical Simulation in Nursing, 5(3), 113-117
- [Background] Abbas, A., Shaltout, A., & Fathalla, M. (2019). The Merit of Simulation in Teaching Medical Interns Vaginal Examination on Laboring Women. American Journal of Obstetrics And Gynecology, 220(1).